CLINICAL TRIAL: NCT00325468
Title: An Open-label, Single-arm Extension Study to Evaluate the Long-term Safety of Denosumab Administration in Postmenopausal Women With Low Bone Mineral Density
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050233
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Low Bone Mineral Density
Keywords: bone loss; osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 162 (Experimental): AMG 162; 60 mg/mL of Denosumab given to all subjects at Screening/Day 1, Month 6, Month 12, Month 18, Month 24, Month 30, Month 36 and Month 42
  Interventions: Drug: AMG 162

INTERVENTIONS:
Drug: AMG 162 — AMG 162; 60 mg/mL of Denosumab given to all subjects at Screening/Day 1, Month 6, Month 12, Month 18, Month 24, Month 30, Month 36 and Month 42

SUMMARY:
An Open-label, Single-arm Extension Study to Evaluate the Long-term Safety of Denosumab Administration in Postmenopausal Women with Low Bone Mineral Density

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ambulatory
* Subject must have atteneded the 20010223 end-of-study visit and have completed all tests and procedures during the end-of-study visit
* signed informed consent must be obtained before any study-specific procedures

Exclusion Criteria:

* Experienced severe and/or serious adverse event which were thought to be related to denosumab administration during the 20010223 study.
* Developed grade 3 or 4 laboratory abnormalities based on Common Terminology Criteria for Adverse Events v3.0 during the 20010223 study which did not normalized upon follow up or did not have diagnosis or treatment.
* Newly diagnosed conditions such as hyper/hypo thyroidism, rheumatoid arthritis, other bone diseases, renal disease.
* Using therapies while participating in the 20010223 study such as oral bisphosphonates, calcitonin, oral strontium, SERMS, systemic glucocortiocosteriods.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2011-03-28 (Actual); Study Completion 2012-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Miller PD, Wagman RB, Peacock M, Lewiecki EM, Bolognese MA, Weinstein RL, Ding B, San Martin J, McClung MR. Effect of denosumab on bone mineral density and biochemical markers of bone turnover: six-year results of a phase 2 clinical trial. J Clin Endocrinol Metab. 2011 Feb;96(2):394-402. doi: 10.1210/jc.2010-1805. Epub 2010 Dec 15. PMID 21159841
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who successfully completed the double-blind, randomized, 4-year dose-ranging parent study 20010223
Groups:
- Placebo: In the parent study 20010223, this cohort received placebo SC for 4 years. Treatment for 4 years in the current study represents initial exposure to denosumab 60 mg Q6M.
- Denosumab 210 mg Q6M: In the parent study 20010223, this cohort received denosumab 210 mg SC Q6M for 2 years and placebo Q6M for 2 years. These subjects were retreated with denosumab 60mg Q6M for 4 years in the current study.
- Denosumab 30 mg Q3M: In the parent study 20010223, this cohort received denosumab 30 mg SC Q3M for 2 years, placebo Q6M for 1 year, followed by denosumab 60 mg Q6M for 1 year. These subjects were treated with denosumab 60 mg Q6M for 4 years in the current study.
- Denosumab Continuous Treatment: In the parent study 20010223, this cohort received denosumab SC for 4 years. During the first 2 years, the doses were 6 mg Q3M, 14 mg Q3M, 14 mg Q6M, 60 mg Q6M, or 100 mg Q6M. During the last two years, all subjects received 60 mg Q6M. Treatment for 4 years in the current study represents 8 years of continuous exposure to denosumab for this cohort.
- Alendronate 70mg QW: In the parent study, this cohort received alendronate 70 mg orally (PO) QW for 2 years; treatment was discontinued for the remaining 2 years of parent Study 20010223. Treatment for 4 year in the current study represents initial exposure to denosumab in subjects previously treated with alendronate.
Period: Overall Study
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW
Started | 23 | 17 | 14 | 124 | 22
Completed | 12 | 12 | 10 | 90 | 14
Not Completed | 11 | 5 | 4 | 34 | 8
Not completed — Adverse Event | 1 | 1 | 0 | 5 | 1
Not completed — Death | 2 | 0 | 2 | 4 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 2
Not completed — Physician Decision | 1 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 14 | 4
Not completed — site closure etc | 4 | 2 | 1 | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW | Total
Number analyzed (Participants) | 23 | 17 | 14 | 124 | 22 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (9.1) | 65.8 (9.4) | 68.0 (7.2) | 65.8 (7.0) | 66.6 (8.9) | 66.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 14 | 124 | 22 | 200
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 18 | 16 | 12 | 112 | 20 | 178
  Black or African American | 0 | 0 | 1 | 2 | 0 | 3
  Hispanic or Latino | 5 | 1 | 1 | 8 | 2 | 17
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Japanese | 0 | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Aborigine | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0
Baseline Bone Mineral Density T-score of Each Anatomic Site [Mean (Standard Deviation); unit: T-score] — A bone mineral density (BMD) T-score is unit-less and represents the difference, in terms of number of standard deviations, between a subject's BMD value and the average BMD value of a gender-specific young normal reference.
  T-score
    Lumbar spine BMD T-score | -2.36 (0.62) | -2.02 (1.16) | -1.29 (0.94) | -1.35 (0.87) | -1.64 (1.09) | -1.55 (0.96)
    Total hip BMD T-score | -1.63 (0.75) | -1.39 (0.67) | -1.05 (0.75) | -1.08 (0.68) | -1.50 (0.81) | -1.21 (0.73)
    Distal 1/3 radius T-score | -1.91 (1.25) | -1.45 (0.98) | -1.14 (1.29) | -1.23 (1.21) | -1.57 (0.98) | -1.35 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Parent Study 20010223 Baseline to Year 8
Time Frame: 8 years
Population: Subjects with nonmissing value at parent study 20010223 baseline and Year 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW
Number analyzed (Participants) | 12 | 12 | 8 | 88 | 13
percent | 8.4 [4.4 to 12.4] | 11.2 [7.2 to 15.2] | 11.0 [6.0 to 16.0] | 16.5 [14.9 to 18.1] | 12.4 [8.5 to 16.4]

2. Secondary Outcome: Bone-Specific Alkaline Phosphatase Percent Change From Parent Study 20010223 Baseline to Year 8
Time Frame: 8 years
Population: Subjects with nonmissing value at parent study 20010223 baseline and Year 8
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW
Number analyzed (Participants) | 12 | 12 | 10 | 90 | 14
percent | -55.8 [-66.7 to -24.4] | -44.7 [-63.6 to -23.8] | -52.5 [-60.4 to -27.1] | -44.4 [-61.9 to -10.2] | -54.2 [-65.1 to -24.9]

3. Primary Outcome: Total Hip Bone Mineral Density Percent Change From Parent Study 20010223 Baseline to Year 8
Time Frame: 8 years
Population: Subjects with nonmissing value at parent study 20010223 baseline and Year 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW
Number analyzed (Participants) | 12 | 12 | 9 | 87 | 13
percent | 1.1 [-1.2 to 3.5] | 4.3 [2.0 to 6.6] | 2.3 [-0.5 to 5.1] | 6.8 [5.8 to 7.7] | 3.4 [1.1 to 5.7]

4. Primary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Parent Study 20010223 Baseline to Year 8
Time Frame: 8 years
Population: Subjects with nonmissing value at parent study 20010223 baseline and Year 8
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW
Number analyzed (Participants) | 11 | 10 | 9 | 87 | 13
percent | -5.2 [-7.4 to -2.9] | 1.4 [-0.9 to 3.8] | 0.6 [-1.9 to 3.1] | 1.3 [0.5 to 2.2] | -2.2 [-4.3 to -0.1]

5. Secondary Outcome: Serum C-Telopeptide Percent Change From Parent Study 20010223 Baseline to Year 8
Time Frame: 8 years
Population: Subjects with nonmissing value at parent study 20010223 baseline and Year 8
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70mg QW
Number analyzed (Participants) | 12 | 13 | 10 | 89 | 13
percent | -66.4 [-90.8 to -27.3] | -72.0 [-84.9 to -57.4] | -48.0 [-87.9 to 26.8] | -64.6 [-77.3 to -2.7] | -49.8 [-82.0 to -45.4]

ADVERSE EVENTS:
Time Frame: 48 months (i.e., 4 years during the 20050233 extension study)
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Placebo | Denosumab 210 mg Q6M | Denosumab 30 mg Q3M | Denosumab Continuous Treatment | Alendronate 70 mg QW | All Participants
Serious Adverse Events (participants affected / at risk) | 3/23 | 3/17 | 5/14 | 31/124 | 3/22 | 45/200
Other Adverse Events (participants affected / at risk) | 18/23 | 15/17 | 13/14 | 106/124 | 19/22 | 171/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Denosumab 210 mg Q6M (N=17) | Denosumab 30 mg Q3M (N=14) | Denosumab Continuous Treatment (N=124) | Alendronate 70 mg QW (N=22) | All Participants (N=200)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 3 | 0 | 3
Performance status decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0 | 4
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 2
Non-Hodgkin's lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Denosumab 210 mg Q6M (N=17) | Denosumab 30 mg Q3M (N=14) | Denosumab Continuous Treatment (N=124) | Alendronate 70 mg QW (N=22) | All Participants (N=200)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 0 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 2 | 1 | 5
Ear congestion (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0 | 2
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 5 | 0 | 7
Hypothyroidism (Endocrine disorders) | 1 | 2 | 0 | 2 | 1 | 6
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 2
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 3 | 1 | 2 | 13 | 3 | 22
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 1 | 2 | 1 | 1 | 6
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 3
Scleral haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 3
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 2 | 6
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 4 | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 1 | 7
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 2 | 6 | 2 | 11
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 1 | 5
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 6 | 1 | 11
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 2 | 7 | 2 | 11
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 2 | 1 | 5
Oedema peripheral (General disorders) | 1 | 0 | 1 | 7 | 0 | 9
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 1 | 3
Bronchitis (Infections and infestations) | 2 | 4 | 3 | 7 | 1 | 17
Fungal oesophagitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 3
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 5
Influenza (Infections and infestations) | 1 | 0 | 1 | 5 | 3 | 10
Localised infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 10 | 2 | 15
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 1 | 18 | 1 | 23
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 9 | 7 | 2 | 24 | 3 | 45
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 15 | 2 | 20
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 8 | 0 | 11
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 1 | 0 | 4
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 9 | 0 | 13
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3 | 0 | 4
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0 | 3
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 7 | 3 | 15
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 3
Chest X-ray abnormal (Investigations) | 0 | 1 | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 3 | 2 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 4 | 20 | 5 | 37
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1 | 14 | 3 | 25
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 6 | 0 | 8
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 0 | 5
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 7 | 1 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 9 | 0 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 2 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 5 | 1 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0 | 14 | 3 | 23
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 2
Trendelenburg's symptom (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 8 | 0 | 11
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 6 | 0 | 8
Headache (Nervous system disorders) | 1 | 0 | 0 | 8 | 1 | 10
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 2 | 0 | 0 | 3 | 0 | 5
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 3
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 4 | 1 | 6
Syncope (Nervous system disorders) | 0 | 1 | 0 | 3 | 0 | 4
Depression (Psychiatric disorders) | 3 | 3 | 0 | 6 | 2 | 14
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 12 | 0 | 14
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 3 | 1 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 1 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 2 | 0 | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 1 | 5
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 3 | 4 | 13 | 3 | 25
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.